CLINICAL TRIAL: NCT02064933
Title: Analysis of Patients Treated for Wiskott-Aldrich Syndrome Since January 1, 1990 (RDCRN PIDTC-6904)
Brief Title: Patients Treated for Wiskott-Aldrich Syndrome (WAS) Since 1990
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Primary Immune Deficiency Treatment Consortium (PIDTC) (Other); Rare Diseases Clinical Research Network (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT RDCRN PIDTC-6904
Record Dates: First submitted 2014-02-13; First posted 2014-02-17 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Wiskott-Aldrich Syndrome
Keywords: Wiskott-Aldrich Syndrome; Hematopoietic Stem Cell Transplantation; Genetic Therapy
MeSH Terms: conditions — Wiskott-Aldrich Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood and tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Retrospective Cohort (Longitudinal Analysis): Participants with WAS treated at consortium centers since 1990 who have received transplant (Stratum A) or gene therapy (Stratum B)
- Prospective Cohort (Longitudinal Analysis): Participants treated at consortium centers since 1990 who will receive transplant (Stratum A) or gene therapy (Stratum B)
- Cross-Sectional Cohort (Cross-sectional Analysis): Living participants with WAS who have received transplant (Stratum A) or gene therapy (Stratum B) at Consortium Centers 1990-Present And >= 2 Years Post-Transplant

SUMMARY:
Wiskott - Aldrich syndrome (WAS) is a rare serious medical condition that causes problems both with the immune system and with easy bruising and bleeding. The immune abnormalities cause patients with WAS to be very susceptible to infections. Depending on the specific type of primary immune deficiency diseases, there are effective treatments, including antibiotics, cellular therapy and gene therapy, but studies of large numbers of patients are needed to determine the full range of causes, natural history, or the best methods of treatment for long term success.

This multicenter study combines retrospective, prospective and cross-sectional analyses of the transplant experiences for patients with WAS who have already received HCT since 1990, or who will undergo Hematopoietic cell transplant (HCT) during the study period. The retrospective and prospective portions of the study will address the impact of a number of pre and post-transplant factors on post-transplant disease correction and ultimate benefit from HCT and the cross-sectional portion of the study will assess the benefit of HCT 2 years post-HCT in consenting surviving patients.

ELIGIBILITY:
Inclusion Criteria:

* WAS participants will be defined as males who have:

  1. thrombocytopenia (< 100K) AND EITHER molecular diagnosis of WAS OR reduced WASP expression; OR
  2. thrombocytopenia (< 100K) AND positive family history consistent with WAS diagnosis; OR
  3. chronic thrombocytopenia (< 100K for minimum of 3 months) AND low mean platelet volume (MPV below normal range for age) AND EITHER recurrent and/or severe infections requiring treatment and/or eczema OR lack of antibody response to polysaccharide antigens or low IgM.
* Longitudinal Analysis (Retrospective and Prospective)

  1. Stratum A. Participants with WAS who have or will Receive HCT

     * Participants with WAS who have received an HCT since January 1, 1990
  2. Stratum B. Participants with WAS who have or will Receive Gene Transfer

     * Participants in which the intention is to treat with gene transfer with autologous modified cells
* Cross-Sectional Analysis (Strata A and B) 1. Participants with WAS who are surviving and at least 2 years after the most recent HCT or gene therapy.

Exclusion Criteria:

* As this is a natural history study, for both the Longitudinal Analysis and the Cross-Sectional Analysis we will not exclude any patients due to race or age who fit the inclusion criteria.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male WAS participants treated at consortium centers Since 1990
Sampling Method: Non-Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2014-02-02 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Longitudinal Analysis: Overall Survival From Time of HCT/Gene Therapy | an expected average of 5 years
  The event analyzed is death from any cause. The time to this event is the time from HCT/gene therapy to death or last follow-up.
Cross-Sectional Analysis: Proportion of Participants Achieving Full T Cell Reconstitution | an expected average of 5 years
  Full T cell reconstitution is defined by all of the following:
  * CD3 cell count within normal range for age.
  * CD4 cell count within normal range for age.
  * CD8 cell count within normal range for age
  * Donor T cell chimerism > 95%
  * Lymphocyte proliferation to PHA. Proliferative responses to PHA within the normal range (at or above the lower limit of normal).
  When possible the proliferation to PHA should be calculated as a percentage of the lower limit of normal controls for that laboratory; alternatively, the lower limit of normal controls for the day may be used
Cross-Sectional Analysis: Proportion of Participants Achieving Full B Cell Reconstitution | an expected average of 5 years
  Full B cell reconstitution is defined by all of the following:
  * Quantitative immunoglobulins (IgG, IgM, and IgA) within normal range; each immunoglobulin level will be assessed separately.
  * Serologic confirmation of post immunization tetanus titer in protective range.
  * Serologic confirmation of post immunization pneumococcal titers in protective range (protective titers for > 50% of the serotypes contained in the vaccine) following immunization
Cross-Sectional Analysis: Proportion of Participants Achieving Resolution of thrombocytopenia | an expected average of 5 years
  Resolution of thrombocytopenia defined by Platelets ≥ 150,000/microliter (transfusion independent for at least 7 consecutive days)
Cross-Sectional Analysis: Day of Recovery of Absolute Neutrophil Count (ANC) to 500 / uL | an expected average of 5 years
  Day of Recovery of Absolute Neutrophil Count (ANC) to 500 / uL is defined as the first day of at least 3 different days the ANC is measured as 500 / uL or greater
Cross-sectional Analysis: Day of Recovery of Platelet Count to 20,000 / uL | an expected average of 5 years
  Day of Recovery of Platelet Count to 20,000 / uL is defined as the first day of at least 3 laboratory values obtained on different days where the platelet count was measured as 20,000 / uL or greater, AND without platelet transfusions for at least 7 consecutive days immediately preceding this day.
Cross-sectional Analysis: Day of Recovery of Platelet Count to 50,000 / uL | an expected average of 5 years
  Day of Recovery of Platelet Count to 50,000 / uL is defined as the first day of at least 3 laboratory values obtained on different days where the platelet count was measured as 50,000 / uL or greater, AND without platelet transfusions for at least 7 consecutive days immediately preceding this day.

SECONDARY OUTCOMES:
Longitudinal Analysis: Proportion of Participants Achieving Hematologic Reconstitution | an expected average of 5 years
  Hematologic Reconstitution is defined as attainment of each of the following lab test values:
  * Hemoglobin within normal range for age
  * WBC count within normal range for age
  * Absolute neutrophil count (ANC) within normal range for age
  * Platelet count ≥ 150,000/microL and without transfusion for at least 7 consecutive days
Longitudinal Analysis: Day of Recovery of Absolute Neutrophil Count (ANC) to 500 / uL | an expected average of 5 years
  Day of Recovery of Absolute Neutrophil Count (ANC) to 500 / uL is defined as the first day of at least 3 different days the ANC is measured as 500 / uL or greater.
Longitudinal Analysis: Day of Recovery of Platelet Count to 20,000 / uL | an expected average of 5 years
  Day of Recovery of Platelet Count to 20,000 / uL is defined as the first day of at least 3 laboratory values obtained on different days where the platelet count was measured as 20,000 / uL or greater, AND without platelet transfusions for at least 7 consecutive days immediately preceding this day.
Longitudinal Analysis: Day of Recovery of Platelet Count to 50,000 / uL | an expected average of 5 years
  Day of Recovery of Platelet Count to 50,000 / uL is defined as the first day of at least 3 laboratory values obtained on different days where the platelet count was measured as 50,000 / uL or greater, AND without platelet transfusions for at least 7 consecutive days immediately preceding this day.
Longitudinal Analysis: Proportion of Participants Achieving Full T Cell Immune Reconstitution | an expected average of 5 years
  * Absolute CD3 T cell count within normal range for age
  * Absolute CD4 T cell count within normal range for age
  * Absolute CD8 T cell count within normal range for age
  * Proliferative responses to PHA within the normal range (at or above the lower limit of normal).
  * When possible the proliferation to PHA should be calculated as a percentage of the lower limit of normal controls for that laboratory; alternatively, the lower limit of normal controls for the day may be used.
Longitudinal Analysis: Proportion of Participants Achieving Full B Cell Immune Reconstitution | an expected average of 5 years
  * Quantitative immunoglobulins (IgG, IgM, and IgA) within normal range for age; each immunoglobulin level will be assessed separately.
  * Serologic confirmation of post immunization tetanus titer in protective range.
  * Serologic confirmation of post immunization pneumococcal titers in protective range (protective titers for > 50% of the serotypes contained in the vaccine) following immunization.
  * Patients who remain on IVIG will be considered not B cell reconstituted.
  * Normalization of isohemagglutinin titers.
Longitudinal Analysis: State of Lineage Specific Chimerism (HCT Stratum) | an expected average of 5 years
  Peripheral blood chimerism will be assessed by FISH XX/XY, STRs, or WASP expression.
Longitudinal Analysis: Definition of Graft Failure / Rejection | an expected average of 5 years
  * Less than 5% of donor cells in all lineages or in whole blood by 100 days post-HCT using standard PCR based or in situ hybridization techniques OR
  * Second transplant by 100 days post-HCT (unless > 5% CD3 and purpose is to boost immune recovery).
  Failure to achieve ≥5% donor cells in all lineages or in whole blood by 100 days post-HCT will be defined as graft failure/rejection. Patients who receive a second transplant by day 100 will be considered graft failure.
Longitudinal Analysis: Severe bleeding episodes | an expected average of 5 years
  Any severe bleeding episode requiring platelet and/or RBC transfusion(s)
Longitudinal Analysis: Malignancy | an expected average of 5 years
  New onset or relapse of lymphoid malignancy confirmed by relevant pathologic and genetic features.
Longitudinal Analysis: Growth | an expected average of 5 years
  Z score of weight and height pre-HCT/gene therapy and post-HCT/gene therapy.
Longitudinal Analysis: Incidence of Acute GVHD | an expected average of 5 years
  The occurrence of skin, gastrointestinal or liver abnormalities fulfilling the Consensus criteria of Grades IIIV or grades III-IV acute GVHD1 are considered events. Death is a competing risk, and patients alive without acute GVHD will be censored at the time of last follow-up.
Longitudinal Analysis: Incidence of Chronic GVHD | an expected average of 5 years
  Chronic GVHD will be graded as limited or extensive.2 Occurrence of symptoms in any organ system that meet the criteria of chronic GVHD will be recorded. Death is a competing risk, and patients alive without chronic GVHD will be censored at time of last follow-up.
Longitudinal Analysis: Autoimmunity disorders | an expected average of 5 years
  Incidence of documented autoimmunity disorders
Longitudinal Analysis: Infections / blood borne infections | an expected average of 5 years
  1. Clinical resolution of any pre-HCT opportunistic infections including but not limited to CMV, HSV1, adenovirus, EBV, and VZV. Approximate time to resolution (clinically well, off treatment, and/or negative culture/PCR assay) will be measured from the day of HCT.
  2. Incidence of documented severe (requiring hospitalization or resulting in death) and/or recurrent bacterial, viral or fungal infection post HCT. These will be reported by site of disease, organism, date of onset post HCT, and whether or not the infection resolved.
  3. Presence and resolution of severe warts (verruca vulgaris, flat warts) from the day of HCT. Whether the subject had complete resolution, partial resolution, persistent or recurrent warts will be recorded.
  4. New episodes of infections due to meningococcus, pneumococcus or hemophilus.
  5. Lymphoproliferative disease due to EBV.
Cross-sectional Analysis: Current State of Lineage Specific Chimerism (HCT Stratum) | an expected average of 5 years
  Peripheral blood donor chimerism will be assessed by FISH XX/XY, STR, and/or WASP expression
Cross-sectional Analysis: Current frequency and severity of infections | an expected average of 5 years
Cross-sectional Analysis: Current Status of Growth | an expected average of 5 years
  Current Z score of weight and height pre-HCT/gene therapy and post-HCT/gene therapy.
Cross-Sectional Analysis: Graft-versus-host Disease (GvHD) | an expected average of 5 years
  Presence of chronic GVHD, current assessment; graded as limited or extensive
Cross-Sectional Analysis: Autoimmunity Disorders | an expected average of 5 years
  Presence of autoimmunity disorders
Cross-sectional Analysis: Severe Bleeding Episodes | an expected average of 5 years
  Any severe bleeding episode requiring platelet and/or RBC transfusion(s) during the previous year.
Cross-sectional Analysis: fertility | an expected average of 5 years
  Whether the subject has biological offspring will be recorded.
Cross-sectional Analysis: malignancy | an expected average of 5 years
  New onset or relapse of lymphoid malignancy confirmed by relevant pathologic and genetic features.
Cross-sectional Analysis: Quality of Life Questionnaire | an expected average of 5 years
  Age appropriate testing will be performed at the cross-sectional visit inpatients surviving at least two years post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: Lauri M. Burroughs, MD, Study Chair — Fred Hutchinson Cancer Center; David J. Rawlings, MD, Study Chair — Department of Pediatrics, University of Washington-Seattle Children's Hospital; Luigi D. Notarangelo, MD, Study Chair — National Institute of Allergy and Infectious Diseases, NIH; Alexandra H. Filipovich, MD, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (43):
- United States (38):
  - Department of Pediatrics, University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Cancer and Blood Disease Institute, Children's Hospital Los Angeles, Keck School of Medicine, University of Southern California, Los Angeles, California
  - Department of Pediatrics, David Geffen School of Medicine at University of California, Los Angeles,, Los Angeles, California
  - Lucile Salter Packard Children's Hospital at Stanford, Palo Alto, California
  - University of California, San Francisco Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Denver, University of Colorado, Denver, Colorado
  - Nemours Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Hospital-George Washington University School of Medicine and Health Sciences, Washington D.C., District of Columbia
  - Blood and Marrow Transplant Program, Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Aflac Cancer and Blood Disorders Center, Emory/Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Center for Cancer and Blood Disorders, Children's Hospital/Louisiana State University, New Orleans, Louisiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Department of Pediatrics, C. S. Mott Children's Hospital, University of Michigan, Ann Arbor, Michigan
  - Division of Pediatric Blood and Marrow Transplantation, University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Children's Center, Rochester, Minnesota
  - Cardinal Glennon Children's Hospital, Saint Louis University, St Louis, Missouri
  - Saint Louis Children's Hospital, Washington University, St Louis, Missouri
  - Institute for Pediatric Cancer and Blood Disorders, Hackensack University Medical Center, Hackensack, New Jersey
  - Department of Pediatrics, Memorial Sloan Kettering Cancer Center, New York, New York
  - Department of Pediatrics, Golisano Children's Hospital, University of Rochester, Rochester, New York
  - Maria Fareri Children's Hospital, New York Medical College, Valhalla, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, University of Cincinnati, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Division of Pediatric Hematology/Oncology, Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Pediatrics, University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine Section of Immunology, Allergy, and Retrovirology, Texas Children's Hospital, Houston, Texas
  - Texas Transplant Institute, Methodist Children's Hospital, San Antonio, Texas
  - Primary Children's Hospital, University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center and University of Washington-Seattle Children's Hospital, Seattle, Washington
  - American Family Children's Hospital, University of Wisconsin, Madison, Wisconsin
  - Children's Hospital of Wisconsin-Milwaukee, Milwaukee, Wisconsin
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Cancer Care Manitoba, University of Manitoba, Winnipeg, Manitoba
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Department of Pediatrics, University of Montreal, Montreal, Quebec

REFERENCES:
- [Background] Griffith LM, Cowan MJ, Kohn DB, Notarangelo LD, Puck JM, Schultz KR, Buckley RH, Eapen M, Kamani NR, O'Reilly RJ, Parkman R, Roifman CM, Sullivan KE, Filipovich AH, Fleisher TA, Shearer WT. Allogeneic hematopoietic cell transplantation for primary immune deficiency diseases: current status and critical needs. J Allergy Clin Immunol. 2008 Dec;122(6):1087-96. doi: 10.1016/j.jaci.2008.09.045. Epub 2008 Nov 6. PMID 18992926
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Kohn DB, Puck JM, Pai SY, Ballard B, Bauer SC, Bleesing JJ, Boyle M, Brower A, Buckley RH, van der Burg M, Burroughs LM, Candotti F, Cant AJ, Chatila T, Cunningham-Rundles C, Dinauer MC, Dvorak CC, Filipovich AH, Fleisher TA, Bobby Gaspar H, Gungor T, Haddad E, Hovermale E, Huang F, Hurley A, Hurley M, Iyengar S, Kang EM, Logan BR, Long-Boyle JR, Malech HL, McGhee SA, Modell F, Modell V, Ochs HD, O'Reilly RJ, Parkman R, Rawlings DJ, Routes JM, Shearer WT, Small TN, Smith H, Sullivan KE, Szabolcs P, Thrasher A, Torgerson TR, Veys P, Weinberg K, Zuniga-Pflucker JC; workshop participants. Primary Immune Deficiency Treatment Consortium (PIDTC) report. J Allergy Clin Immunol. 2014 Feb;133(2):335-47. doi: 10.1016/j.jaci.2013.07.052. Epub 2013 Oct 15. PMID 24139498
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Kohn DB, Puck JM, Shearer WT, Burroughs LM, Torgerson TR, Decaluwe H, Haddad E; workshop participants. Primary Immune Deficiency Treatment Consortium (PIDTC) update. J Allergy Clin Immunol. 2016 Aug;138(2):375-85. doi: 10.1016/j.jaci.2016.01.051. Epub 2016 Apr 22. PMID 27262745
- [Result] Pai SY, Logan BR, Griffith LM, Buckley RH, Parrott RE, Dvorak CC, Kapoor N, Hanson IC, Filipovich AH, Jyonouchi S, Sullivan KE, Small TN, Burroughs L, Skoda-Smith S, Haight AE, Grizzle A, Pulsipher MA, Chan KW, Fuleihan RL, Haddad E, Loechelt B, Aquino VM, Gillio A, Davis J, Knutsen A, Smith AR, Moore TB, Schroeder ML, Goldman FD, Connelly JA, Porteus MH, Xiang Q, Shearer WT, Fleisher TA, Kohn DB, Puck JM, Notarangelo LD, Cowan MJ, O'Reilly RJ. Transplantation outcomes for severe combined immunodeficiency, 2000-2009. N Engl J Med. 2014 Jul 31;371(5):434-46. doi: 10.1056/NEJMoa1401177. PMID 25075835
- [Result] Haddad E, Allakhverdi Z, Griffith LM, Cowan MJ, Notarangelo LD. Survey on retransplantation criteria for patients with severe combined immunodeficiency. J Allergy Clin Immunol. 2014 Feb;133(2):597-9. doi: 10.1016/j.jaci.2013.10.022. Epub 2013 Dec 10. No abstract available. PMID 24331379
- [Result] Shearer WT, Dunn E, Notarangelo LD, Dvorak CC, Puck JM, Logan BR, Griffith LM, Kohn DB, O'Reilly RJ, Fleisher TA, Pai SY, Martinez CA, Buckley RH, Cowan MJ. Establishing diagnostic criteria for severe combined immunodeficiency disease (SCID), leaky SCID, and Omenn syndrome: the Primary Immune Deficiency Treatment Consortium experience. J Allergy Clin Immunol. 2014 Apr;133(4):1092-8. doi: 10.1016/j.jaci.2013.09.044. Epub 2013 Nov 28. PMID 24290292
- [Result] Dvorak CC, Cowan MJ, Logan BR, Notarangelo LD, Griffith LM, Puck JM, Kohn DB, Shearer WT, O'Reilly RJ, Fleisher TA, Pai SY, Hanson IC, Pulsipher MA, Fuleihan R, Filipovich A, Goldman F, Kapoor N, Small T, Smith A, Chan KW, Cuvelier G, Heimall J, Knutsen A, Loechelt B, Moore T, Buckley RH. The natural history of children with severe combined immunodeficiency: baseline features of the first fifty patients of the primary immune deficiency treatment consortium prospective study 6901. J Clin Immunol. 2013 Oct;33(7):1156-64. doi: 10.1007/s10875-013-9917-y. Epub 2013 Jul 2. PMID 23818196
- [Result] Griffith LM, Cowan MJ, Notarangelo LD, Puck JM, Buckley RH, Candotti F, Conley ME, Fleisher TA, Gaspar HB, Kohn DB, Ochs HD, O'Reilly RJ, Rizzo JD, Roifman CM, Small TN, Shearer WT; Workshop Participants. Improving cellular therapy for primary immune deficiency diseases: recognition, diagnosis, and management. J Allergy Clin Immunol. 2009 Dec;124(6):1152-60.e12. doi: 10.1016/j.jaci.2009.10.022. PMID 20004776
- [Result] Burroughs LM, Petrovic A, Brazauskas R, Liu X, Griffith LM, Ochs HD, Bleesing JJ, Edwards S, Dvorak CC, Chaudhury S, Prockop SE, Quinones R, Goldman FD, Quigg TC, Chandrakasan S, Smith AR, Parikh S, Davila Saldana BJ, Thakar MS, Phelan R, Shenoy S, Forbes LR, Martinez C, Chellapandian D, Shereck E, Miller HK, Kapoor N, Barnum JL, Chong H, Shyr DC, Chen K, Abu-Arja R, Shah AJ, Weinacht KG, Moore TB, Joshi A, DeSantes KB, Gillio AP, Cuvelier GDE, Keller MD, Rozmus J, Torgerson T, Pulsipher MA, Haddad E, Sullivan KE, Logan BR, Kohn DB, Puck JM, Notarangelo LD, Pai SY, Rawlings DJ, Cowan MJ. Excellent outcomes following hematopoietic cell transplantation for Wiskott-Aldrich syndrome: a PIDTC report. Blood. 2020 Jun 4;135(23):2094-2105. doi: 10.1182/blood.2019002939. PMID 32268350
- [Derived] Alexander JL, Davila Saldana BJ, Brazauskas R, Dammalapati SG, Griffith LM, Shah AJ, Shimano KA, Ochs HD, Bleesing J, Ebens CL, Kapadia M, Bauchat A, Kapoor N, Oved JH, Eissa H, Lust H, Keller MD, Haines H, Chandrakasan S, Talano JM, Rayes A, Madden LM, Shereck EB, Miller HK, Forbes Satter LR, Martinez CA, Rozmus J, Bednarski JJ, Yu LC, Chellapandian D, Aquino VM, Knutsen AP, Chong H, Chopek A, Gillio AP, Joshi A, Rangarajan HG, Moore TB, Andolina JR, DeSantes K, Vander Lugt MT, Prockop SE, Shyr D, Sullivan KE, Parikh SH, Weinacht KG, Torgerson TR, Marsh RA, Dvorak CC, Chan AY, Haddad E, Heimall J, Pulsipher MA, Leiding JW, Kohn DB, Puck JM, Notarangelo LD, Rawlings DJ, Cowan MJ, Petrovic A, Pai SY, Burroughs LM. Hematopoietic Cell Transplantation for Wiskott-Aldrich syndrome: A PIDTC Report. Blood Adv. 2025 Dec 4:bloodadvances.2025017662. doi: 10.1182/bloodadvances.2025017662. Online ahead of print. PMID 41346295
- See also: Primary Immune Deficiency Treatment Consortium (PIDTC), Rare Clinical Diseases Research Network, National Institutes of Health — https://www.rarediseasesnetwork.org/cms/pidtc/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/